CLINICAL TRIAL: NCT00926991
Title: Chest Wall Stabilization for Traumatic Chest Wall Injuries: An Observational Study
Brief Title: Chest Wall Repair of Rib Fractures After Trauma
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Jose J. Diaz, Jr., MD, Vanderbilt University Medical Center
Other Study IDs: Acute chest wall injuries
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- traumatic rib fractures
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention; observation only

SUMMARY:
This is a prospective, observational trial of 50 patients who have multiple, severe rib fractures following trauma. The investigators will follow their hospital stay for outcomes (infections, length of stay and medical care) as well as their early post-hospital course.

DETAILED DESCRIPTION:
Hypothesis:

Rib fracture repair utilizing open reduction and internal fixation with commercially available rib plating systems improves outcomes (i.e., infectious complications), decreases hospital stay and mortality.

Study Design:

This is a prospective, observational study of 50 patients who, due to their injury pattern, are operative candidates for open reduction and internal fixation with commercial available rib plating systems for one of the following indications:

1. Flail chest with/without failure to wean from the ventilator
2. Significantly displaced rib fractures with/without lung impalement
3. Symptomatic multiple rib fractures - Failure of pain control

Outcome measures to be evaluated include:

1. Hospital Mortality
2. Ventilator free days
3. Need for tracheotomy
4. Infectious Complications (pneumonia, bacteremia, UTI, empyema)
5. Hospital & ICU Days
6. Disposition following discharge

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least >18 years of age
* Subjects must have one of the following clinical indications:
* >3 rib flail segments with paradoxical chest wall movement
* Non-repair of defect may result in pulmonary hernia
* Minimal associated injuries
* Severely displaced fractures are significantly impeding lung expansion.
* Failure of narcotics or epidural pain catheter to control pain

Exclusion Criteria:

* Significant pulmonary contusion
* Significant brain injury (AIS 4 and/or ICP monitoring)
* Severe associated injuries which, in the opinion of the surgeon will preclude operative chest wall stabilization
* Subjects not expected to survive the 90-day follow-up period
* Known pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vanderbilt University Trauma Center.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
pain scales | daily
ventilator requirement | daily
hospital days | discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Diaz, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States